CLINICAL TRIAL: NCT02729337
Title: Affecting the Epidemiology of HIV in Uganda Through Older Adolescents
Brief Title: Affecting the Epidemiology of HIV in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Innovative Public Health Research (Other)
Collaborators: Internet Solutions for Kids Uganda (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MH109296
Record Dates: First submitted 2016-03-15; First posted 2016-04-06 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Sexual Abstinence; HIV; Contraceptive Usage
Keywords: technology; adolescent; developing country; hiv prevention; mHealth
MeSH Terms: conditions — Sexual Abstinence; Contraception Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ITG (In This Together) (Experimental): This will be a multi-week behavioral intervention delivered daily via text messaging. Content will be based upon the IMB model of HIV preventive behavior and informed by our formative work.
  Interventions: Behavioral: ITG (In This Together)
- Control Group (No Intervention): Given the preliminary nature of the intervention development, the control group will be inactive but blinded. They will receive two messages per week encouraging them to make healthy sexual decisions to reduce their HIV risk. Messages will be didactic and not driven by the IMB model.

INTERVENTIONS:
Behavioral: ITG (In This Together) — Comprehensive, mHealth-based HIV prevention program for Ugandan adolescents 18-22 years of age.
  Arms: ITG (In This Together)

SUMMARY:
The investigators propose to develop a comprehensive, text messaging-based HIV prevention program for Ugandan adolescents 18-22 years of age.

DETAILED DESCRIPTION:
The investigators propose to develop a comprehensive, text messaging-based HIV prevention program for Ugandan adolescents 18-22 years of age. The guiding theoretical model is the Information-Motivation-Behavioral Skills (IMB) Model of HIV Preventive Behavior.

Intervention development will be iterative: In Phase 1, the investigators will identify an intervention content "map." Then, online focus groups (FG) will be conduct online with Ugandan young adults (n = 40-80) to confirm program components (e.g., social support via Text Buddy, optimal time of delivery of daily text messages) and saliency of intended program topics.

In Phase 2, the investigation team will "translate" content into a bank of text messages that will be reviewed for comprehensiveness and inclusion of the most pertinent topics. The final pool of messages among Ugandan young adults will be tested in the Content Advisory Council (CAC; n = 30) to assess their reactions to the content, scope, style, and tone of the messages.

In Phase 3, the investigators will merge the content with the software program developed to deliver the intervention and then internally conduct a functionality test of the programmed messages. Following, the protocol and program will be tested in a beta test of 20 Ugandan adults.

In Phase 4, the investigators will test the intervention in a randomized controlled trial of 200 Ugandan young adults randomly assigned to either the intervention (n = 100) or control (n = 100) arms. The main outcome measures will focus on feasibility (e.g., recruitment and retention rates) and acceptability (e.g., Text Buddy). The primary efficacy outcome measures, measured at 3-months post-intervention, will be: (a) frequency of unprotected sex acts; (b) sustained sexual abstinence, and (c) increased HIV testing rates.

Specific Aims are as follows:

Specific Aim 1: Design a 6-week text messaging-based HIV prevention and healthy sexuality program for adolescents 18-22 years old.

Specific Aim 2: Pilot test the intervention for feasibility and acceptability among 18- to 22-year-old Ugandans.

Specific Aim 3: Obtain preliminary data needed for a larger-scale controlled trial services study to examine program efficacy.

ELIGIBILITY:
Inclusion Criteria:

* living in Uganda
* aged 18-22 years
* able to read English
* exclusive owner of a cell phone
* using text messaging for at least 6 months
* intended to have the same phone number or the next six months
* able to access the Internet (to complete online surveys)
* able to provide informed consent

Exclusion Criteria:

* no other exclusion criteria will be applied

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Program feasibility: Recruitment | 24 weeks
  The number of participants recruited for the RCT (n=200)
Program feasibility: Retention | Through study completion, an average of 6 weeks
  The number of participants that will remain in the study at program end (80%)
Program acceptability as assessed by a scale created for the RCT | At intervention end, 6-weeks post baseline
  Participant ratings of program features (e.g., Text Buddy) at intervention end

SECONDARY OUTCOMES:
Percent of participants reporting condom use during sex as assessed by self-report | At intervention end, 6-weeks post baseline
  The percent of participants who report, at intervention end, using condoms during sex always versus not using condoms at least once, during the intervention period
Percent of participants reporting abstinence as assessed by self-report | At intervention end, 6-weeks post baseline
  The percent of participants who report, at intervention end, not having sex versus having sex at least once, during the intervention period
Percent of participants who have gotten an HIV test as assessed by self-report | At intervention end, 6-weeks post baseline
  The percent of participants who report, at intervention end, having gotten an HIV test versus not, during the intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Michele Ybarra, MPH PHD, Principal Investigator — Center for Innovative Public Health Research
Locations (1):
- Internet Solutions for Kids Uganda, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ybarra ML, Agaba E, Nyemara N. A Pilot RCT Evaluating InThistoGether, an mHealth HIV Prevention Program for Ugandan Youth. AIDS Behav. 2021 Oct;25(10):3437-3448. doi: 10.1007/s10461-021-03237-5. Epub 2021 May 7. PMID 33963477

DOCUMENTS (1):
  • Informed Consent Form (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT02729337/ICF_000.pdf